CLINICAL TRIAL: NCT00160303
Title: Prolotherapy vs. Corticosteroid Therapy for the Treatment of Lateral Epicondylitis of the Elbow, A Randomized Controlled Trial.
Brief Title: Efficacy Study of Prolotherapy vs Corticosteroid for Tennis Elbow
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 04-1561; 2005P-001080
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Lateral Epicondylitis
Keywords: Prolotherapy; Lateral Epicondylitis; Tennis Elbow; Corticosteroid Therapy
MeSH Terms: conditions — Tennis Elbow | interventions — Prolotherapy

INTERVENTIONS:
Drug: Prolotherapy
Drug: Local Corticosteroid Therapy

SUMMARY:
The purpose of the research is to study the effects of two different injection therapies for the treatment of lateral epicondylitis (tennis elbow). Specifically, we will look at which therapy provides better short and long-term relief of pain, which treatment allows better function and less disability, and which treatment gives back better strength in the affected hand. Each subject will receive only one of the two treatments. Although both of these treatments are usually very well tolerated, it is important to make this comparison because it is believed that one of these therapies may have better long term effectiveness, with a lower cost, and smaller number of potential side effects.

DETAILED DESCRIPTION:
Lateral Epicondylitis or tennis elbow is one of the most commonly diagnosed upper-extremity musculoskeletal disorders seen in general practice. It is characterized by painful enthesopathy or tendinosis of the common extensor tendon at the outer region of the elbow at the fibro-osseous junction. "Although tennis elbow" was originally made note of in the medical literature by Runge in 1873, the term derives from "Lawn Tennis Arm" later described by Morris in 1882.

Traditionally, lateral epicondylitis causes characteristic pain in the lateral elbow region and is often associated with significant morbidity. It occurs most commonly in individuals between 40 and 50 years and equally affects both men and women. The dominant arm is involved in 75% of patients. While other etiologies have been proposed, including radial nerve entrapment, it is generally agreed that tennis elbow is the result of repetitive mechanical micro-trauma and overuse, but many cases have no biomechanical association, nor vocational or avocational correlation. This condition is often brought about by repeated flexion and extension of the wrist or by a direct injury to the epicondyle or elbow. However, most patients are unable to recall or to identify a precipitating event. The average duration of an episode of lateral epicondylitis is 6 to 24 months, and 10% to 30% of cases result in work absenteeism, leading to a high loss of productivity. Numerous treatment options have been described for lateral epicondylitis. Most cases are managed in primary care settings, and although there are more than forty possible treatments, there is still a lack of consensus about optimal therapeutic management. Moreover, most of these treatments lack sound scientific evidence.

The preferred method of treatment of lateral epicondylitis often involves corticosteroid injections with or without the addition of local anesthetic. In general, injection of local corticosteroids is commonly used to reduce inflammation in patients with chronic tendinopathies such as lateral epicondylitis. However, since inflammation is not necessarily a major feature in this lesion, and if present, may present a vital component of the healing response. Inhibiting this process may result in a suboptimal outcome. Thereby, despite their popularity, the rationale for use of corticosteroids is controversial and the evidence for long-term benefit lacks. Likewise, potential side effects such as infection, tissue atrophy, pigmentation changes, hyperglycemia, etc. do exist. Moreover, many of the recommendations for the use of corticosteroid injections are anecdotal. In a review by Labelle et al, it was concluded that there was insufficient scientific evidence to support the use of corticosteroids injections for lateral epicondylitis. Assendelft et al came to similar conclusions in his review when he found that existing evidence on corticosteroid injections for lateral epicondylitis was unclear and that questions regarding the optimal timing, dosage, injection, technique, and injection volume remained unanswered.

Prolotherapy, though not as yet extensively studied, is another emerging therapy presenting as an alternative to corticosteroid injection for the treatment of lateral epicondylitis. It continues to rise in popularity, especially by clinicians who commonly treat musculoskeletal injuries. With its early origins dating back to the time of Hippocrates, prolotherapy is defined as the iatrogenic stimulation of wound healing and tissue repair process through the injection of an irritant solution into damaged ligaments, tendons, and joints thus encouraging their healing and repair.

Essentially, this occurs as a result of a localized inflammatory reaction with stimulation of rounds cell infiltration with resultant collagen synthesis, and formation of firm permanent fibrous tissue and bone. The new collagen runs parallel to existing ligaments and tendons and has a linear orientation, resulting in ultimate strengthening and stabilization of the ligament, tendon, or joint with subsequent reduction of pain. It is generally safe and very well tolerated and has been used throughout the western medical community for over 50 years.

Existing research on prolotherapy began in the 1930s when Lerich first described the rich supply of nerve endings in articular ligaments. This was re-introduced by Gardner in 1953. Also in the 1950s, Hackett, who described most joint pain as ligamentous, was the first to scientifically demonstrate a method of strengthening ligaments by injection of a proliferant solution. At that time, the use of an irritant solution was thought to work by creation of a scar tissue rather than by development of a proliferative response. As pain was perceived to arise when normal tension on a ligament stretched the relaxed ligament fibers, which resulted in abnormal tension and stimulation of the sensory nerves because the nerve fibers did not stretch, reduction of pain was thereby thought to arise with stabilization of these relaxed ligaments through generation of a strong scar tissue about that structure. Reduction of pain was realized by Hackett who reported an 82% success rate in the treatment of chronic spinal pain in 1816 patients treated during a 20-year period.

A subsequent study in 1982 on rabbit ligaments by Lui et al showed that prolotherapy might have a positive effect on mass, thickness, enthesis strength, and weight-to-length ratio of injected ligaments, as compared to controls. A different study by Klein et al in 1989 showed histological documentation of ligament proliferation in human subjects. This was in response to proliferative injections, which objectively increased the diameter of collagen fibers with an associated decrease in pain as well as an objective increase in range of motion. In another study, Ongley et al found a statistically significant reduction in ligamentous laxity 9 months after injecting the ends of collateral and cruciate ligaments of knees that had substantial ligamentous laxity as measured by a computerized knee analysis device. All of these studies found decreases in pain levels of patients involved.

In addition to early studies, which focused on the mechano-proliferative effects, later studies in proliferant injection therapy considered its affect on both subjective pain levels and more objective outcomes such as functional status. For example, in Ongley's study, more patients in the experimental group showed improvements in pain with a concomitant decrease in levels of disability. Faber et al, using a dextrose, phenol, and glycerin containing proliferant, were able to document an increase in the size of sacroiliac ligaments. They also were able to show a moderate to marked improvement in pain and function in subjects who received prolotherapy in concert with manipulation versus controls who received saline injections and sham manipulations. Reeves et al showed that prolotherapy solution consisting of 10% dextrose resulted in clinically and statistically significant improvements in patients with knee osteoarthritis. The clinically significant changes were seen in joint pain, subjective joint swelling, flexion range of motion, and in tendency to buckle, all signs which significantly impact level of function.

Although these and other studies have shown positive effects of proliferant therapy on mechanical properties of ligaments as well as subjective improvements in pain and function, most have suffered from small sample size, inadequate controls, and inconsistency of study design and methodology. Kim et al reviewed and critically analyzed three randomized, controlled studies on the use of dextrose, glycerin, and phenol prolotherapy for chronic low back pain. They found inconclusive data to support its use due to the lack of adequate controls, heterogeneity in patient diagnoses, and variations in solutions injected. Nevertheless, clinical use of prolotherapy warrants further investigation.

As lateral epicondylitis involves a cascade of injury at or about the insertion of the common extensor tendon at the fibro-osseous junction, the patho-physiologic response to proliferation at this joint seems promising. Based on previous studies, prolotherapy would theoretically strengthen and stabilize the overstretched and torn strands of fibrous tissue that cause the cascade of instability and generation of pain at this junction. Not only would prolotherapy thereby improve subjective pain, it would improve objective strength and stability of the joint with resultant increase in function. Moreover, in doing so, prolotherapy would benefit both the patient and society at large by offering a relatively safer, less expensive, and longer lasting alternative to corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* age criteria >18yo, <75yo, history of pain > 3 months, < 2 years; pain on resisted extension of wrist and/or middle finger test, (resisted extension of middle finger at the MCP joint)
* local tenderness to palpation at the lateral epicondyle
* subject can read and write in English.

Exclusion Criteria:

* history of steroid injections within 6 months prior to intervention;
* other arm/forearm pathology such as radial nerve compression; pregnancy/nursing;
* known thrombocytopenia, coagulopathy, or bleeding diathesis; history of diffuse pain syndrome;
* history of Inflammatory Arthropathy;
* Workman's Compensation (RSI) > 2 years; patients with litigation pending/planned; patients who are unable to return for F/U;
* intolerance/allergy to local anesthetics or injection corticosteroids; fear of needles; untreated depression;
* history of narcotic use for pain management greater than 1 month or history of narcotic abuse problem.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2005-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
10 cm Visual Analogue Scale (VAS)
Disabilities of the Arm, Shoulder, and Hand (DASH)

SECONDARY OUTCOMES:
Grip Strength

CONTACTS AND LOCATIONS:
Overall Officials: Joanne P Borg-Stein, MD, Principal Investigator — Spaulding Rehabilitation Hospital; Alexios G Carayannopoulos, DO, MPH, Study Director — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Wellesley Outpatient Center, Wellesley, Massachusetts, United States